CLINICAL TRIAL: NCT04354311
Title: Relationship Between the ANI Score During Standardized Painful Stimulation and the Nociceptive Response to Laryngoscopy Intubation
Brief Title: Prediction of Hemodynamic Response to Intubation by ANI Variation During Standardized Stimulation
Acronym: ANI_LARYNGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012_34; 2013-A01127-38 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2020-04

CONDITIONS: Tracheal Intubation Morbidity; Pain
Keywords: ANI; hemodynamic responses; tracheal intubation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, analytical, monocentric, piloted study
Masking Description: Patients under general anesthesia during the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Anesthetic induction : total target-controlled intravenous anesthesia d was used with propofol and remifentanil. The effect site was then gradually increased to obtain a satisfaction depth of anesthesia. Assisted ventilation was then started by facemask ventilation (Sat O2>95% and expired CO2 fraction normal, tidal volume of 8 mL/kg, a respiratory rate of 12 cycles per minute, with an FiO2 100% with no positive end expiratory pressure.
  After stabilisation period of 2 minutes and record of the patient's parameters, a standardized nociceptive stimulation was applied at the level of the ulnar nerve (PTC of 50 Hz at 70 mA). The variation of ANI score and hemodynamic parameters were collected during the 2 following minutes.
  After stabilization of ANI, orotracheal intubation was attempted. Maximal variation of heart rate (HR), blood pressure and the occurrence of somatic manifestations (intense cough, movement, tears) were recorded.
  Interventions: Device: ANI

INTERVENTIONS:
Device: ANI — Under steady state total intravenous anaesthesia with propofol and remifentanil at constant dosage, tetanus stimulation of the ulnar nerve was performed followed by orotracheal intubation. The variation of ANI and hemodynamic parameters as well as the somatic response associated with both maneuvers were collected.

SUMMARY:
The objective : to investigate a correlation between ANI following a standardized nociceptive stimulus and hemodynamic or somatic reactions during orotracheal intubation.

Piloted study. ANI and hemodynamic and somatic parameters response associated tetanus stimulation followed by orotracheal intubation were collected.

DETAILED DESCRIPTION:
Background: The Analgesia Nociception Index reflects the balance between analgesia and nociception and allows early detection of a defect in analgesia. Orotracheal intubation is responsible for a sometimes deleterious hemodynamic reaction. The Analgesia Nociception Index could allow an individual adjustment of the investigator's anesthetic inductions during this period.

Objective: The objective of this study is to investigate if there is a correlation between variations in the ANI following a standardized nociceptive stimulus and the occurrence of hemodynamic or somatic reactions during orotracheal intubation without muscle relaxation.

Materials and Methods: Prospective, interventional, analytical, monocentric, piloted study carried out in the operating theatre after obtaining patient's informed consent between January 2014 and November 2014. Under steady state total intravenous anaesthesia with propofol and remifentanil at constant dosage (entropy between 40 and 60) tetanus stimulation of the ulnar nerve was performed followed by orotracheal intubation. The variation of ANI and hemodynamic parameters as well as the somatic response associated with both maneuvers were collected.

ELIGIBILITY:
Inclusion Criteria:

* Any patient requiring general anaesthesia with tracheal intubation by direct laryngoscopy
* Intubation Difficulty Assessment Score < 7
* BMI between 17 and 30 Kg/m2
* Socially insured patient
* Patient 18 years of age or older
* Patient with signed consent
* Patient with a sinus heart rhythm

Exclusion Criteria:

* Patient refusing to participate in the study
* Pregnant woman
* Patient with a pace maker (any mode)
* Patient treated with Beta Blocker
* Known Dysautonomia
* Diabetes
* Spontaneous ventilation anaesthesia
* Allergy to any of the required medications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
predictability of hemodynamic impact during laryngoscopy by tetanus-induced ANI variation, | measurement during intubation, an average 40 seconds and 5 minutes
  area under the corresponding Receiver Operating Characteristic curve with DeltaTetanus as dependent variable, and Hemodynamic Impact as state variable

SECONDARY OUTCOMES:
predictability of somatic impact during laryngoscopy by tetanus-induced ANI variation, | observation during intubation, an average between 40 seconds and 5 minutes
  area under the corresponding Receiver Operating Characteristic curve with DeltaTetanus as dependent variable, and Somatic Impact as state

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Jozefowicz, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France

REFERENCES:
- [Result] Jozefowicz E, Sabourdin N, Fontaine V, Lambelin V, Lejeune V, Menu H, Bourai M, Tavernier B. Prediction of reactivity during tracheal intubation by pre-laryngoscopy tetanus-induced ANI variation. J Clin Monit Comput. 2022 Feb;36(1):93-101. doi: 10.1007/s10877-020-00624-6. Epub 2021 Jan 2. PMID 33387153